CLINICAL TRIAL: NCT02653820
Title: Complementary Effect of Reflexology on Chemotherapy-Induced Nausea and Vomiting
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 102-15 HYMC
Record Dates: First submitted 2016-01-06; First posted 2016-01-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Reflexology
MeSH Terms: interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy patients (Experimental): Chemotherapy patients will receive reflexology treatment
  Interventions: Other: Reflexology

INTERVENTIONS:
Other: Reflexology

SUMMARY:
Reflexology treatment may influence the severity of chemotherapy-induced nausea and vomiting. This study aims to investigate the clinical effect of reflexology on chemotherapy-induced nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Chemotherapy patients

Exclusion Criteria:

* Myocardial Infarction in previous 6 months
* Mechanical colonic obstruction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Change in Severity of Nausea | Three weeks
  Nausea will be assessed both before after three weeks of reflexology treatment by Common Toxicity Criteria Adverse Events Tool
Change in Severity of Vomiting | Three weeks
  Vomiting will be assessed both before after three weeks of reflexology treatment by Common Toxicity Criteria Adverse Events Tool

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Shulman, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No